CLINICAL TRIAL: NCT00607750
Title: A Phase 2 Randomized, Double-Masked, Study to Evaluate the Safety and Preliminary Efficacy of ATG003 in Patients With Neovascular Age-Related Macular Degeneration (NV-AMD) Receiving Frequent Maintenance Intravitreal Anti-VEGF Antibody Therapy (Ranibizumab or Bevacizumab)
Brief Title: Safety and Efficacy of ATG003 in Patients With AMD Receiving Anti-VEGF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CoMentis (Industry)
Responsible Party: Carl Grove, President, CoMentis, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATG003-203
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2010-10

CONDITIONS: Age-Related Macular Degeneration
Keywords: Wet AMD, Comentis, ATG003, mecamylamine
MeSH Terms: conditions — Macular Degeneration | interventions — Mecamylamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- ATG003 (Experimental)
  Interventions: Drug: ATG003 (mecamylamine)

INTERVENTIONS:
Drug: ATG003 (mecamylamine) — 1% Ophthalmic solution, eyedrop BID, 48 weeks
  Arms: ATG003
Drug: Placebo — Placebo eyedrops, BID, 48 weeks
  Arms: 1

SUMMARY:
This study is a double-masked, randomized, placebo-controlled study of the safety and preliminary efficacy of ATG003 (topical mecamylamine) in patients receiving maintenance injections of either ranibizumab or bevacizumab. Study Hypothesis: Mecamylamine could be effective in the treatment of neovascular AMD.

ELIGIBILITY:
Inclusion Criteria:

* > 55 years of age
* clinical diagnosis of neovascular AMD

Exclusion Criteria:

* confounding ocular condition

Min Age: 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-05; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of ATG003 (mecamylamine HCL ophthalmic solution) | Day 1 - Week 50

SECONDARY OUTCOMES:
To evaluate the efficacy of ATG003 | Day 1 - Week 50

CONTACTS AND LOCATIONS:
Overall Officials: Carl Grove, MS, Study Director — Comentis, Inc.